CLINICAL TRIAL: NCT02294357
Title: A Phase 2 Study of Weekly 70 mg/m2 Carfilzomib for Multiple Myeloma Patients Refractory to 27 mg/m2 Carfilzomib
Brief Title: Weekly 70 mg/m2 Carfilzomib for Multiple Myeloma Patients Refractory to 27 mg/m2 Carfilzomib
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to the difficulties to enroll subjects.
Sponsor: Oncotherapeutics (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IST-CAR-2014-100701 (20159897)
Record Dates: First submitted 2014-11-10; First posted 2014-11-19 (Estimated); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: Multiple Myeloma
Keywords: carfilzomib; proteasome inhibitor; multiple myeloma; relapsed/refractory
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — carfilzomib; Dexamethasone; Calcium Dobesilate; dexamethasone acetate; Prednisone; Methylprednisolone; Methylprednisolone Acetate; Lenalidomide; pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Carfilzomib + Dexamethasone (Experimental): Carfilzomib will be administered at 70 mg/m2 as an infusion over 30 minutes on days 1, 8 and 15 of a 28-day cycle. Dexamethasone (IV or PO) will be given prior to each carfilzomib administration.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone
- Carfilzomib + Prednisone (Experimental): Carfilzomib will be administered at 70 mg/m2 as an infusion over 30 minutes on days 1, 8 and 15 of a 28-day cycle. Prednisone (IV or PO) will be given prior to each carfilzomib administration.
  Interventions: Drug: Carfilzomib; Drug: Prednisone
- Carfilzomib + Methylprednisolone (Experimental): Carfilzomib will be administered at 70 mg/m2 as an infusion over 30 minutes on days 1, 8 and 15 of a 28-day cycle. Methylprednisolone(IV or PO) will be given prior to each carfilzomib administration.
  Interventions: Drug: Carfilzomib; Drug: Methylprednisolone
- Carfilzomib+Lenalidomide+Dexamethasone (Experimental): Carfilzomib will be administered at 70 mg/m2 as an infusion over 30 minutes on days 1, 8 and 15 of a 28-day cycle. Dexamethasone (IV or PO) will be given prior to each carfilzomib administration. Lenalidomide will be given at the same dose and schedule as patient was receiving previously.
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Lenalidomide
- Carfilzomib+Pomalidomide+Dexamethasone (Experimental): Carfilzomib will be administered at 70 mg/m2 as an infusion over 30 minutes on days 1, 8 and 15 of a 28-day cycle. Dexamethasone (IV or PO) will be given prior to each carfilzomib administration. Pomalidomide will be given PO at 4mg daily on days 1-21 of a 28-day cycle
  Interventions: Drug: Carfilzomib; Drug: Dexamethasone; Drug: Pomalidomide

INTERVENTIONS:
Drug: Carfilzomib
  Other Names: Kyprolis
Drug: Dexamethasone — If the patient was receiving steroids at the equivalent of > 8 mg of dexamethasone weekly either intravenously (IV) or Per Orem (PO) in combination with carfilzomib, the same drug(s), dose(s) and schedule(s) of steroids will be continued. If the patient was not receiving steroids or was receiving less than the equivalent of 8 mg of dexamethasone weekly, then he/she will be given 8 mg of dexamethasone (IV or PO) prior to each carfilzomib administration.
  Other Names: Decadron; Dexamethasone acetate
  Arms: Carfilzomib + Dexamethasone; Carfilzomib+Lenalidomide+Dexamethasone; Carfilzomib+Pomalidomide+Dexamethasone
Drug: Prednisone — f the patient was receiving prednisone, at the equivalent of > 8 mg of dexamethasone weekly PO in combination with carfilzomib, he/she will continue to receive prednisone at the same dose and schedule.
  Other Names: Deltasone; Cortan
  Arms: Carfilzomib + Prednisone
Drug: Methylprednisolone — If the patient was receiving methylprednisolone at the equivalent of > 8 mg of dexamethasone weekly either IV or PO in combination with carfilzomib, he/she will continue to receive methylprednisolone at the same dose and schedule.
  Other Names: Medrol; Methylprednisolone acetate
  Arms: Carfilzomib + Methylprednisolone
Drug: Lenalidomide — given at same dose and schedule as patient was receiving while being treated with twice weekly carfilzomib at 27 mg/m2
  Other Names: Revlimid
  Arms: Carfilzomib+Lenalidomide+Dexamethasone
Drug: Pomalidomide — administered PO at 4mg daily on days 1-21 of a 28 day cycle
  Other Names: Pomalyst
  Arms: Carfilzomib+Pomalidomide+Dexamethasone

SUMMARY:
The purpose of this Phase II study is to evaluate the safety and effectiveness (good and bad effects) of carfilzomib given as a 30-minute infusion and at a dose of 70 mg/m2 to treat patients with multiple myeloma (MM), who are currently showing progressive disease (worsening) and had progressed (did not respond to treatment) within 8 weeks of receiving treatment with twice weekly 27mg/m2 of carfilzomib. Carfilzomib is approved by the U.S. Food and Drug Administration (FDA) to be used only in certain U.S. patients with relapsed and refractory multiple myeloma that have tried and failed other therapies. Carfilzomib is considered an investigational drug for this study because the dose and regimen included in this study are different from the FDA approved carfilzomib regimen. Carfilzomib is a type of drug called a proteasome inhibitor. Carfilzomib is thought to work by preventing breakdown of abnormal proteins in cells, causing the cells to die. Cancer cells are more sensitive to these effects than normal cells. Carfilzomib has been previously given to more than 1800 people in clinical trials.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open label, non-randomized study to evaluate the safety and efficacy of a 30-minute infusion of 70 mg/m2 of carfilzomib among MM patients who are currently showing progressive disease (PD) and had failed their last treatment with twice weekly 27mg/m2 of carfilzomib alone or as part of a combination regimen.

The study will consist of 1) a screening period; 2) up to eight 28-day, treatment cycles; 3) maintenance treatment; 4) a final assessment to occur 28 days after the end of the last treatment cycle; and 5) a follow-up period. The study will enroll a total of 45 patients who are currently showing PD and had progressed within 8 weeks of receiving their last treatment with twice weekly 27mg/m2 of carfilzomib alone or as part of a combination regimen. Additionally, patients who have not achieved a complete response (CR) and have plateaued (as defined by unchanged disease markers for at least 8 weeks) while treated with a combination of carfilzomib (twice weekly 27 mg/m2), lenalidomide and dexamethasone; carfilzomib (twice weekly 27 mg/m2), pomalidomide and dexamethasone; or carfilzomib (twice weekly 27 mg/m2) and dexamethasone are also eligible for this study. Patients who were treated with a carfilzomib (twice weekly 27 mg/m2) containing combination who are currently on carfilzomib (twice weekly 27 mg/m2) and dexamethasone with or without lenalidomide or pomalidomide maintenance therapy and are not in CR and show unchanged disease markers for at least 8 weeks will also be eligible.

Patients will be enrolled from 15 hematology/oncology sites across the United States.

During the treatment period, all doses of carfilzomib will be given at 70 mg/m2 infused over 30 minutes. Among patients who received steroids at the equivalent of > 8 mg of dexamethasone weekly with carfilzomib, steroids will be administered using the same drug(s) at the same dose(s) and schedule(s) as they received during their previous carfilzomib treatment. Patients who did not receive steroids or received the equivalent of less than 8 mg of dexamethasone weekly will be given 8 mg of dexamethasone prior to each carfilzomib administration. Carfilzomib will be administered at a facility capable of managing hypersensitivity reactions. Pre- and post-dose intravenous (IV) hydration (between 250 mL and 500 mL normal saline or other appropriate IV fluid formulation) may be given at the discretion of the treating physician. Subjects should be monitored periodically during this period for evidence of fluid overload. Subjects who complete 8 cycles without showing PD will be eligible to receive maintenance therapy on a 28-day cycle with carfilzomib and steroids as administered during the last cycle of the treatment period. In addition, those treated with lenalidomide with carfilzomib and dexamethasone will continue lenalidomide at the same dose and schedule as used during the treatment period. For those treated with pomalidomide with carfilzomib and dexamethasone, pomalidomide will be administered at the same dose and schedule as during treatment.

During maintenance (cycle 9 and beyond), carfilzomib will be administered at the dose received during the last cycle of study treatment on Days 1, 8 and 15, and steroids will be administered using the same drug(s) at the same dose(s) and schedule(s) as given during the last cycle of study treatment. Patients will remain on maintenance therapy until documentation of PD as defined by the modified Bladé criteria or until they develop toxicity. Patients with stable disease (SD) will remain on maintenance therapy. Dose reductions of carfilzomib and steroids will be permitted as per protocol guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. Has a diagnosis of MM based on standard criteria as follows:

   Major criteria:
   * Plasmacytomas on tissue biopsy.
   * Bone marrow plasmacytosis (greater than 30% plasma cells).
   * Monoclonal immunoglobulin (Ig) spike on serum electrophoresis IgG greater than 3.5 g/dL or IgA greater than 2.0 g/dL; kappa or lambda light chain excretion greater than 1 g/day on 24-hour urine protein electrophoresis.

   Minor criteria:
   * bone marrow plasmacytosis (10% to 30% plasma cells)
   * monoclonal immunoglobulin present but of lesser magnitude than given under major criteria
   * lytic bone lesions
   * normal IgM less than 50 mg/dL, IgA less than 100 mg/dL, or IgG less than 600 mg/dL

   Any of the following sets of criteria will confirm the diagnosis of multiple myeloma:
   * any 2 of the major criteria
   * major criterion 1 plus minor criterion 2, 3, or 4
   * major criterion 3 plus minor criterion 1 or 3
   * minor criteria 1, 2, and 3, or 1, 2, and 4
2. Patient must meet one of the following:

   * Currently, patient has progressive MM that has progressed while receiving twice weekly carfilzomib 27mg/m2 alone or as part of their last carfilzomib-containing combination regimen
   * Currently, the patient is not in CR and plateaued (as defined by unchanged disease markers for at least 8 weeks) while treated with carfilzomib (twice weekly 27 mg/m2) and dexamethasone with or without lenalidomide or pomalidomide
   * Patients who were previously receiving a carfilzomib (twice weekly 27 mg/m2) containing regimen and are currently receiving carfilzomib (twice weekly 27mg/m2) and dexamethasone maintenance therapy with or without lenalidomide or pomalidomide and are not in CR and have plateaued
3. Patient must have received at least one full cycle of carfilzomib at a dose of twice weekly 27mg/m2 prior to showing evidence of PD or plateauing from their last carfilzomib-containing regimen.
4. Patient must have previously received treatment with an immunomodulatory agents lenalidomide or pomalidomide to be eligible for the study (applicable only for subjects who qualify via inclusion criteria 2B or 2C).
5. There is no limit to the number of prior lines of therapy that a patient may have received.
6. Measurable disease, as defined by one or more of the following (assessed within 14 days prior to first dose):

   * Serum M-protein ≥ 0.5 g/dL, or
   * Urine M-protein ≥ 200 mg/24 hours, or
   * Only in patients who do not meet a or b, then use serum free light chain (SFLC) > 100 mg/L (involved light chain) and an abnormal κ/λ ratio
7. Age ≥ 18 years.
8. Life expectancy ≥ 6 months.
9. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
10. Adequate hepatic function within 14 days prior to first dose, with bilirubin < 1.5 × the upper limit of normal (ULN), and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 3 × ULN.
11. LVEF ≥ 40%. 2-D transthoracic echocardiogram (ECHO) is the preferred method of evaluation. Multigated Acquisition Scan (MUGA) is acceptable if ECHO is not available.
12. Absolute neutrophil count (ANC) ≥ 1000/mm3 within 14 days prior to first dose. Screening ANC is to be independent of granulocyte colony stimulating factor support for ≥ 1 week and pegylated granulocyte colony stimulating factor for ≥ 2 weeks.
13. Hemoglobin ≥ 8.0 g/dL within 14 days prior to enrollment. Use of erythropoietic stimulating factors and red blood cell (RBC) transfusions per institutional guidelines is allowed; however, most recent RBC transfusion must have been at least 7 days prior to obtaining screening hemoglobin.
14. Platelet count ≥ 75,000/mm3 (≥ 50,000/mm3 if myeloma involvement in the bone marrow is > 50%) within 14 days prior to first dose. Patients must not have received platelet transfusions for at least 7 days prior to obtaining the screening platelet count.
15. Calculated or measured creatinine clearance (CrCl) of ≥ 30 mL/min within 14 days prior to first dose. Calculations are based on a standard formula, such as the Cockcroft and Gault: [(140 - Age) × Mass (kg) / (72 × Creatinine mg/ dL)]; multiply result by 0.85 if female.
16. Written informed consent in accordance with federal, local, and institutional guidelines.
17. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within the 7 days prior to study drug administration and a negative urine pregnancy test within the 3 days prior to the first study drug administration
18. WOCBP and male subjects who are sexually active with WOCBP must agree to use 2 highly effective methods of contraception during the study and for 30 days following the last dose of study treatment including a male condom.

Exclusion Criteria:

1. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
2. Plasma cell leukemia (> 2.0 × 109/L circulating plasma cells by standard differential)
3. Waldenström's macroglobulinemia
4. Amyloidosis
5. Glucocorticoid therapy (prednisone > 30 mg/day or equivalent) within 7 days prior to first dose
6. Cytotoxic chemotherapy with approved or investigational anticancer therapeutics within 28 days prior to first dose
7. Treatment with bortezomib (Velcade®), thalidomide, pomalidomide (Pomalyst®) or lenalidomide (Revlimid®) within 21 days prior to first dose
8. Focal radiation therapy within 7 days prior to first dose. Radiation therapy to an extended field involving a significant volume of bone marrow within 21 days prior to enrollment (i.e., prior radiation must have been to < 30% of the bone marrow)
9. Immunotherapy within 21 days prior to first dose
10. Major surgery within 21 days prior to first dose
11. Active congestive heart failure (New York Heart Association [NYHA] Classes III to IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention. Myocardial infarction within 6 months prior to first dose. Echocardiogram or MUGA evidence of left ventricular ejection fraction (LVEF) below institutional normal within 28 days prior to enrollment
12. Acute active infection requiring systemic antibiotics, antiviral (except antiviral therapy directed at HBV), or antifungal agents within 14 days prior to first dose
13. Known human immunodeficiency virus (HIV) seropositivity
14. Known active hepatitis B or C virus infection (except for patients with HBV receiving and responding to HBV antiviral therapy: these patients are allowed)
15. Patients with known cirrhosis
16. Second malignancy within the past 3 years, except:

    * Adequately treated basal cell or squamous cell skin cancer
    * Carcinoma in situ of the cervix
    * Prostate cancer < Gleason score 6 with stable prostate-specific antigen (PSA) over 12 months
    * Breast carcinoma in situ with full surgical resection
    * Treated medullary or papillary thyroid cancer
17. Patients with myelodysplastic syndrome
18. Significant neuropathy (Grades 3 to 4) within 14 days prior to first dose
19. Peripheral neuropathy with pain ≥ G2 within 14 days prior to first dose
20. Patients with baseline hepatic impairment
21. Women who are pregnant and/or breast feeding
22. Known hypersensitivity to dexamethasone
23. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
24. Hypersensitivity to any of the required concomitant drugs or supportive treatments, including hypersensitivity to antiviral drugs.
25. Prior participation in any Onyx-sponsored Phase 3 trial
26. Ongoing graft-versus-host disease
27. Pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to enrollment
28. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to enrollment
29. Any other clinically significant medical disease or psychiatric condition that, in the Investigator's opinion, may interfere with protocol adherence or a patient's ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2014-12; Primary Completion 2020-09-21 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | up to 30 months
  Complete response (CR)+ very good partial response (VGPR) + partial response (PR), defined using International Myeloma Working Group (IMWG) criteria
Clinical Benefit Rate (CBR) | up to 30 months
  CBR=ORR + minor response (MR)
Number of patients undergoing adverse events | up to 36 months
  Adverse events (AEs) graded via the Common Terminology Criteria for Adverse Events (CTCAE) v4.03 criteria

SECONDARY OUTCOMES:
Time to Progression (TTP) | 36 months
  Time from initiation of therapy to progressive disease
Progression-Free Survival (PFS) | 36 months
  Time from initiation of therapy to progressive disease or death from any cause, whichever occurs first
Time to Response (TTR) | 36 months
  Time from the initiation of therapy to the first evidence of a confirmed response
Duration of Response (DOR) | 36 months
  Time from the first response (> PR) to progressive disease
Overall Survival (OS) | 36 months
  Time from initiation of therapy to death from any cause or last follow-up visit

CONTACTS AND LOCATIONS:
Overall Officials: James R Berenson, MD, Principal Investigator — James R. Berenson MD, Inc.
Locations (7):
- United States (7):
  - California Cancer Associates for Research & Excellence (cCARE), Encinitas, California
  - Wellness Oncology and Hematology, West Hills, California
  - James R Berenson, MD, Inc., West Hollywood, California
  - Cancer Specialists of North Florida, Fleming Island, Florida
  - Hudson Valley Hem/Onc Associates, Poughkeepsie, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Blood & Cancer Center of East Texas, Tyler, Texas

IPD SHARING:
Plan to Share IPD: No
Demographics and Clinical Responses